CLINICAL TRIAL: NCT04562909
Title: Evaluation of Postural Control in Premature Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2020.815
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Premature Birth
Keywords: premature; postural control; balance
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premature children: Premature children born before than 32 weeks were included.
  Interventions: Device: Neurocom balance master device
- Healthy Control Group: Age matched healthy controls
  Interventions: Device: Neurocom balance master device

INTERVENTIONS:
Device: Neurocom balance master device — With the Modified Sensory Balance Interaction Clinical Test, the static balance will be examined by measuring the torso oscillation velocities while the eyes are open and the eyes closed on the stable rigid and unstable foam floors, and the dynamic balance will be examined with the sit-stand test, which is the basic motor activity in daily life, and the parameters will be measured on the same device.

SUMMARY:
To date, it is largely unknown whether preterm children experience balance problems and whether they have normal postural control. Assuming that postural adaptation is affected after preterm delivery because it depends on attention and fine motor control, the postural control and motor development of children born preterm less than 32 weeks in the 5-7 age period will be affected compared to their healthy controls. Identifying these situations according to their healthy peers will improve the general health of premature births and enable better intervention methods to be designed.

DETAILED DESCRIPTION:
Thanks to modern technical interventions and trained health personnel, the survival rate of premature babies has increased significantly in recent years. Neurodevelopmental abnormalities increase as birth weight and gestational week decrease and the presence of adverse biological conditions add up. Brain structures involved in fine motor control, such as the cerebellum, basal ganglia, corpus callosum, amygdala, and hippocampus, are smaller in babies born preterm, even without premature brain damage. Many of the problems associated with these in children are often difficult to detect at an early age, so numerous symptoms may not be detected until school age. In this sense, making periodic assessments of the progress in each child's motor development is essential to identifying deficiencies and thus facilitates referral to early intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Premature children born less than 32 weeks
* Age between 5-7 years
* Neurological development to be normal
* Giving an informed consent

Exclusion Criteria:

* Not giving an informed consent

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature and healthy children
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
Neurocom balance master | Day 0
  With the Modified Sensory Balance Interaction Clinical Test, the static balance will be examined by measuring the torso oscillation velocities while the eyes are open and the eyes closed on the stable rigid and unstable foam floors, and the dynamic balance will be examined with the sit-stand test, which is the basic motor activity in daily life, and the parameters will be measured on the same device.

CONTACTS AND LOCATIONS:
Overall Officials: Naime Evrim Karadag-Saygi, Prof, Study Director — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aylward GP. Neurodevelopmental outcomes of infants born prematurely. J Dev Behav Pediatr. 2014 Jul-Aug;35(6):394-407. doi: 10.1097/01.DBP.0000452240.39511.d4. PMID 25007063
- [Background] Stoinska B, Gadzinowski J. Neurological and developmental disabilities in ELBW and VLBW: follow-up at 2 years of age. J Perinatol. 2011 Feb;31(2):137-42. doi: 10.1038/jp.2010.75. Epub 2010 Jul 15. PMID 20634795
- [Background] Brandt T, Schautzer F, Hamilton DA, Bruning R, Markowitsch HJ, Kalla R, Darlington C, Smith P, Strupp M. Vestibular loss causes hippocampal atrophy and impaired spatial memory in humans. Brain. 2005 Nov;128(Pt 11):2732-41. doi: 10.1093/brain/awh617. Epub 2005 Sep 1. PMID 16141283
- [Background] Allin M, Matsumoto H, Santhouse AM, Nosarti C, AlAsady MH, Stewart AL, Rifkin L, Murray RM. Cognitive and motor function and the size of the cerebellum in adolescents born very pre-term. Brain. 2001 Jan;124(Pt 1):60-6. doi: 10.1093/brain/124.1.60. PMID 11133787